CLINICAL TRIAL: NCT00072527
Title: Induction Cisplatin/Irinotecan Followed By Combination Carboplatin, Etoposide And Chest Radiotherapy In Limited Stage Small Cell Lung Cancer: A Phase II Study
Brief Title: Cisplatin and Irinotecan Followed by Carboplatin, Etoposide, and Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30206; U10CA031946 (NIH); CDR0000339871 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Cisplatin; Etoposide; Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction and consolidation chemotherapy (Experimental): Induction chemotherapy (Cycles 1 and 2): Patients receive cisplatin 30 mg/m^2 on days 1, 8, 22 and 29 and irinotecan 65 mg/m^2 on days 1, 8, 22 and 29 for cycles 1 and 2.
  Consolidation chemotherapy (Cycles 3, 4 and 5 beginning on day 43, week 7): Patients receive carboplatin on days 43, 64 and 85, etoposide 100 mg/m^2 IV on days 43-45, 64-66 and 85-87 and XRT 5 fractions/week starting on day 43
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: etoposide; Drug: irinotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — IV
Drug: cisplatin — IV
Drug: etoposide — IV
Drug: irinotecan hydrochloride — IV
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, irinotecan, carboplatin, and etoposide, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cisplatin and irinotecan followed by carboplatin, etoposide, and radiation therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of cisplatin and irinotecan followed by carboplatin, etoposide, and radiotherapy, in terms of 2-year survival, in patients with limited stage small cell lung cancer.

Secondary

* Determine the overall response rate, overall survival, and failure-free survival of patients treated with this regimen.
* Determine the response rate in patients treated with induction therapy comprising irinotecan and cisplatin.
* Determine the toxicity and tolerability of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive cisplatin IV over 60 minutes and irinotecan IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
* Consolidation therapy: Immediately after the completion of induction therapy, patients receive carboplatin IV over 60 minutes on day 1 and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Radiotherapy: Beginning on day 1 of consolidation therapy, patients undergo chest radiotherapy daily 5 days a week for 6-7 weeks.

After the completion of consolidation therapy, patients who achieve a complete remission or very good partial remission may undergo prophylactic radiotherapy to the brain.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study within 15-24 months.

ELIGIBILITY:
1. Histologically or cytologically documented small cell lung cancer of limited stage.

   1.1 Limited stage disease category includes patients with disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal lymph nodes.

   1.2 Although they are usually defined as having limited stage small cell lung cancer, because of concern about the volume of the radiation field that would be required, patients with clinically suspected or confirmed supraclavicular lymph node metastases, patients with pathologically enlarged contralateral hilar lymph nodes, and patients with pleural effusions that are visible on plain chest radiographs, whether cytologically positive or not, are NOT eligible.
2. All Patients must have Measurable Disease

   2.1 Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan.

   2.2 Pleural/pericardial effusions are not considered measurable.
3. Age ≥18
4. ECOG Performance status 0-2.
5. Prior Treatment - No prior chemotherapy or radiotherapy for SCLC.
6. No "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.
7. Non-pregnant and non-nursing because of significant risk to the fetus/infant.
8. Required Initial Laboratory Values

   * Granulocytes ≥1,500/µl
   * Platelets ≥100,000/µl
   * Serum Creatinine ≤ULN
   * Bilirubin <1.5 mg/dl
   * SGOT (AST) <2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2003-11; Primary Completion 2007-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Efficacy, in terms of survival, at 2 years after initiation of study treatment

SECONDARY OUTCOMES:
Overall response rate as measured by RECIST at completion of study treatment
Overall survival
Failure-free survival
Response rate as measured by RECIST after completion of 2 courses of induction chemotherapy
Toxicity as measured by NCI CTCAE v.30 after completion of 2 courses of chemotherapy
Tolerability as measured by chemotherapy dose-delivered dose delays after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Kelley, MD, Study Chair — Duke University
Locations (76):
- United States (76):
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center - Plymouth Campus, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Hudner Oncology Center at Saint Anne's Hospital, Fall River, Massachusetts
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Frisbie Memorial Hospital, Rochester, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Gaston Memorial, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Comprehensive Cancer Center at Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Result] Kelley MJ, Bogart JA, Hodgson LD, Ansari RH, Atkins JN, Pang H, Green MR, Vokes EE. Phase II study of induction cisplatin and irinotecan followed by concurrent carboplatin, etoposide, and thoracic radiotherapy for limited-stage small-cell lung cancer, CALGB 30206. J Thorac Oncol. 2013 Jan;8(1):102-8. doi: 10.1097/JTO.0b013e31827628e1. PMID 23196276